CLINICAL TRIAL: NCT02875717
Title: Influence of Acetylsalicylic Acid and Low Molecular Weight Heparins on the Incidence of Renal Hematoma of Shockwave Lithotripsy
Status: Completed | Type: Observational
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Principal Investigator, Christoph Schregel, Resident, Kantonsspital Winterthur KSW
Other Study IDs: 2015-0662/PB_2016-00897
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Urolithiasis; Renal Hematoma
MeSH Terms: conditions — Urolithiasis | interventions — Aspirin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control
- Acetylsalicylic acid: Patients that were on medication with Acetylsalicylic acid on the date of shockwave lithotripsy
  Interventions: Drug: Acetylsalicylic acid
- Low Molecular weight heparin: Patients that were on medication with low molecular heparin on the date of shockwave lithotripsy
  Interventions: Drug: low molecular weight heparin

INTERVENTIONS:
Drug: Acetylsalicylic acid
  Groups: Acetylsalicylic acid
Drug: low molecular weight heparin
  Groups: Low Molecular weight heparin

SUMMARY:
Retrospective Analysis of patients that received shockwave lithotripsy as Treatment of ureteral or kidney Stones. Condition examinated is the effect of low molecular weight Heparins and acetylsalicylic acid on the Formation of renal hematoma after shockwave lithotripsy. Primary outcome is documented hematoma in a postoperative ultrasound control. Secondary outcomes are perioperative complication, Need for erythrocyte tranfusion, interventions for bleeding control, readmission or death within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* consent
* Stones in kidney and proximal Ureter
* Treatment with shockwave lithotripsy for urolithiasis between January 2009 and September 2015 at Kantonsspital Winterthur

Exclusion Criteria:

* other Position of ureteral Stones
* missing data in Patient reports
* refused consent
* under Age limit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that received shockwave lithotripsy at Kantonsspital Winterthur between January 2009 and September 2015 and were 18 years or older at the time of treatment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Renal Hematoma in ultrasound control | first day after intervention

SECONDARY OUTCOMES:
Intervention for bleeding control | 30 days after intervention
Need for erythrocyte concentrate tranfusion | 30 days after intervention
Death | 30 days after intervention
Hospital readmission | 30 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hubert John, M.D., Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterhur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schregel C, John H, Randazzo M, Keller I. Influence of acetylsalicylic acid and low-molecular weight heparins on the formation of renal hematoma after shock wave lithotripsy. World J Urol. 2017 Dec;35(12):1939-1946. doi: 10.1007/s00345-017-2070-0. Epub 2017 Jul 12. PMID 28702844